CLINICAL TRIAL: NCT00736905
Title: Pharmacokinetics, Safety and Tolerability of TMC278 in Subjects With Mildly or Moderately Impaired Hepatic Function
Brief Title: TMC278-TiDP6-C130: Pharmacokinetics, Safety and Tolerability of TMC278 in Subjects With Mildly or Moderately Impaired Hepatic Function.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CR007465
Record Dates: First submitted 2008-08-14; First posted 2008-08-18 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: HIV; AIDS; Hepatic Impairment
Keywords: TMC278-TiDP6-C130; TMC278-C130; healthy volunteer; hepatic impairment; HIV Infections
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Rilpivirine

INTERVENTIONS:
Drug: TMC278

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics (how the drug is absorbed into the bloodstream, distributed in the body and eliminated from the body) after a single dose and after repeated administration of TMC278 administered once daily for 11 days in subjects with mild or moderate hepatic impairment (impaired liver function), compared with healthy control subjects. Furthermore the short-term safety and tolerability (how well the body tolerates the drug) of TMC278 will be assessed.

DETAILED DESCRIPTION:
Human immunodeficiency virus (HIV)-infected patients are routinely being treated with combinations of 3 or 4 drugs (highly active antiretroviral therapy [HAART]), to reduce the risk of viral resistance development. Development of new potent antiretroviral (ARV) drugs is urgently needed to prolong suppression of viral replication in subjects infected with HIV. This is a Phase I, open-label, parallel, controlled, sequential study to investigate the single-dose and steady-state pharmacokinetics, and short-term safety and tolerability of TMC278 in subjects with mild or moderate hepatic impairment compared to subjects with normal hepatic function. The trial aims to provide guidance on administration and dose recommendations of TMC278 in subjects with mildly or moderately impaired hepatic function. The study population will consist of a total of 32 male and female subjects between 18 and 65 years. Panel A will consist of 8 subjects with mild hepatic impairment and 8 healthy subjects matched for sex, age (± 5 yrs), and BMI (± 15%). Panel B will consist of 8 subjects with moderate hepatic impairment and 8 healthy subjects matched for sex, age (± 5 yrs), and BMI (± 15%). Treatment in Panel A and Panel B will be conducted sequentially. Subjects in Panel A will receive a TMC278 25 mg tablet once daily for a total of 11 days. Recruitment for subjects for Panel B will start after evaluation of the safety, tolerability and pharmacokinetic data from subjects in Panel A. The anticipated dose of TMC278 to be administered to subjects in Panel B is the same dose as for Panel A (25 mg once daily for 11 days), but this dose might be adjusted depending on the results of Panel A.

ELIGIBILITY:
Inclusion Criteria:

* Non smoking or smoking no more than 10 cigarettes, or 2 cigars, or 2 pipes per day for at least 3 months prior to selection
* Body Mass Index (BMI, weight in kg divided by the square of height in meters) of 18.0 to 32.0 kg/m2, extremes included
* Only for subjects with hepatic impairment: History of hepatic disease
* Documented liver cirrhosis
* Mild or moderate liver function impairment
* Only for healthy control subjects: Healthy on the basis of a physical examination, medical history, electrocardiogram (ECG), vital signs and the results of blood biochemistry and hematology tests and a urinalysis
* Matched to a subject with hepatic impairment with regards to sex, age (± 5 yrs), and BMI (± 15%).

Exclusion Criteria:

* No positive HIV test
* No females, except if postmenopausal since more than 2 years, or posthysterectomy, or post tubal ligation
* No barbiturate, amphetamine, recreational or narcotic drug use
* No use of more than 1 unit of alcoholic beverages per day
* No positive urine drug test
* No active gastrointestinal disease (with the exception of liver cirrhosis in the hepatically impaired subjects), cardiovascular, neurologic, psychiatric, metabolic, renal, respiratory, inflammatory, or infectious disease
* No currently significant diarrhea, gastric stasis, or constipation
* No history of any significant skin disease
* No previously demonstrated clinically significant allergy or hypersensitivity to any of the excipients of the investigational medication administered in this trial (i.e. TMC278)
* Not previously participated in more than 1 trial with TMC125, TMC120 and/or TMC278 or having developed a rash, erythema or urticaria while participating in a trial with the aforementioned compounds
* No participation in an investigational drug trial within 60 days prior to the first administration of trial medication
* No donation of blood or plasma or significant blood loss within the 60 days preceding the first administration of trial medication
* No vulnerable subjects
* No subjects who are not able to read or write
* Only for subjects with hepatic impairment: No acute or active hepatitis
* No evidence of hepatic decompensation
* No grade 3 or 4 encephalopathy
* No hepatic carcinoma
* No hepatorenal syndrome
* No severe liver insufficiency
* Not an active candidate for liver transplantation
* No grade 3 laboratory abnormalities present with the exception of laboratory abnormalities related to hepatic impairment
* Only for healthy control subjects: No hepatitis A, B or C infection
* No current hepatic disease
* No subjects with certain lab abnormalities.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-06; Primary Completion 2009-09 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to assess the single-dose and steady-state pharmacokinetics of TMC278 in subjects with mild or moderate hepatic impairment compared to matched healthy control subjects.

SECONDARY OUTCOMES:
The secondary objective of this study is to assess the short-term safety and tolerability of TMC278 in subjects with mild or moderate hepatic impairment compared to matched healthy control subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited